CLINICAL TRIAL: NCT05496244
Title: ROBYN Study - Robotic Assisted Surgery in Gynecological Indications Compared to Conventional Laparoscopy - A Prospective, Non-Interventional, Multinational, Post-Market Clinical Investigation
Brief Title: ROBYN Study - Robotic Assisted Surgery in Gynecological Indications Compared to Conventional Laparoscopy
Acronym: ROBYN
Status: Withdrawn | Type: Observational
Why Stopped: Overall re-assessment of study design
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: 1.0
Record Dates: First submitted 2022-07-13; First posted 2022-08-11 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: GYN Disorders
MeSH Terms: conditions — Genital Diseases, Female | interventions — Laparoscopy; Robotic Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Epidemiological Section: Consecutive enrollment of patients with indications of interest
- Observational Section: Extended data collection on patients treated via conventional laparoscopy or robotic-assisted surgery
  Interventions: Device: Laparoscopy; Device: Robotic-assisted surgery

INTERVENTIONS:
Device: Laparoscopy — Laparoscopic surgery
  Groups: Observational Section
Device: Robotic-assisted surgery — Robotic-assisted surgery
  Groups: Observational Section

SUMMARY:
Robotic Assisted Surgery (da Vinci System) in gynecological indications compared to conventional laparoscopy

DETAILED DESCRIPTION:
A Prospective, Non-Interventional, Multinational, Post-Market Clinical Investigation

ELIGIBILITY:
Key Inclusion Criteria:

* Patient is willing to participate and to comply with the study procedures
* Patient present with gynecological disease that may be treated with surgical intervention

Key Exclusion Criteria:

* Life expectancy for less than 1 year

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients present with gynecological disease that may be treated by surgical intervention
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Describe treatment decision | Enrollment Completion
  Describe treatment decision for the procedure of choice
Describe patient outcome | 12 Months
  Describe patient outcome from robotic-assisted surgery and conventional laparoscopy by using physiological parameter such as relief or improvement of symptoms, number of complications or number of re-operations and changes in the patient reported quality of life (EQ-5D-5L) between baseline and FU at 12 Months (changes in the score)
Describe impact of patient factors on outcome | 12 Months
  Describe impact of patient factors on outcome by using physiological parameter, such as age, BMI, uterus size, report co-morbidities
Complications of medical interest | 90 days
  Describe complication of medical interest

SECONDARY OUTCOMES:
Quality of Life Impact per patient reported questionnaires | 12 Months
  Describe Quality of Life impact as assessed via patient reported questionnaires; changes in quality of life questionnaires scores between baseline and up to follow-up 12 months will be assessed (EQ-5D-5L on mobility, self-care, usual activities, pain/discomfort, anxiety/depression)
Describe the impact of surgeon experience on outcome | 12 Months
  Describe the impact of surgeon experience on outcome; individual surgeon experience will be collected (self-reported by surgeon) and linked to every performed procedure; descriptive assessment if the reported surgeon experience has an impact on the outcome, e.g. number of reported complications. As surgeon experience, the number of performed procedures per indication and technique (robotic-assisted surgery or laparoscopy will be collected), as well as the overall years the surgeon is performing surgeries.
Describe the performance and use of Intuitive instruments | 12 Months
  Describe the performance and use of Intuitive instruments; information on any device failure or device deficiency will be collected and descriptively assessed
Describe the performance and use of Intuitive systems | 12 Months
  Describe the performance and use of Intuitive systems; information on any device failure or device deficiency will be collected and descriptively assessed

CONTACTS AND LOCATIONS:
Overall Officials: Ingolf Juhasz-Böss, Prof. Dr., Principal Investigator — Universitätsklinikum Freiburg, Germany; Vincent Lavoué, Prof. Dr., Principal Investigator — CHU de Rennes, France